CLINICAL TRIAL: NCT02055612
Title: Mobile Clinic- a Cross-sectional Epidemiological Survey to Investigate the Prevalence of Wet Aged-related Macular Degeneration (wAMD) in Elderly Population in Slovak Republic
Brief Title: Mobile Clinic - a Cross-sectional Epidemiological Survey
Status: Completed | Type: Observational
Sponsor: Novartis Slovakia, s.r.o. (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRFB002ASK01 EPI
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Age Related Macular Degeneration
Keywords: wet AMD; epidemiology
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to find out prevalence of aged-related macular degeneration (AMD) in Slovak Republic. The outcome of the project will be epidemiology survey, prevalence of wet form of AMD in relation to demographic data, patient´s anamnesis, nutrition, co-morbidities etc.

DETAILED DESCRIPTION:
It´s cross-sectional epidemiological survey, multi-centric, non-interventional

1. Patients will fill a questionnaire with demography data, anamnesis, risk factors.
2. Patients will be assessed by using Amsler grid.
3. Patient´s back of the eye will be examined with fundus camera (searching for long-term back of the eye changes, retina vessels, macula and surrounding tissues) by retina specialist.
4. Patient undergoes optical coherent tomography (OCT) examination (cross-section of fovea and macula) by retina specialist.

The project actively screen patients with wAMD. All patients will sign an informed consent.

The process of screening will be held in certain timeframe (cca. 2 months) and selected areas of Slovak Republic.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (aged≥55 years) from selected areas in Slovak Republic
2. Patients with home base far than 35 km from the nearest center (centers: Bratislava, Nitra, Nové Zámky, Trenčín, Bojnice, Žilina, Martin, Ružomberok, Banská Bystrica, Zvolen, Poprad, Prešov, Košice, Trebišov)
3. Patient´s informed consent signed.

Exclusion Criteria:

* Patients who do not meet the inclusion criteria

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults from general population across Slovak Republic over 55 years of age, predominantly with home base far than 35 km from nearest retina center
Sampling Method: Probability Sample
Enrollment: 3278 (Actual)
Dates: Start 2013-03; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Aged specific prevalence of aged-related macular degeneration | participants screened each day 8 hours during a 2 months period in selected areas according to protocol criteria

SECONDARY OUTCOMES:
Social-demography structure of patients with wAMD | participants screened each day 8 hours during a 2 months period in selected areas according to protocol criteria
Risk factors associated with wAMD (e.g. co-morbidities, nutrition effects) | participants screened each day 8 hours during a 2 months period in selected areas according to protocol criteria
Relation between home distance of the patients with wAMD from the nearest center and availability of heath care | participants screened each day 8 hours during a 2 months period in selected areas according to protocol criteria
Other eye diseases during screening process | participants screened each day 8 hours during a 2 months period in selected areas according to protocol criteria

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Krasnik, M.D., PhD., Principal Investigator — Ophthalmology Clinic of Faculty of Medicine of Comenius University and Bratislava University Hospital
Locations (1):
- Novartis Slovakia, s.r.o., Bratislava, Slovakia